CLINICAL TRIAL: NCT01148186
Title: The Patient as a Driver of Change: an Intervention Study to Reduce the Use and Impact of Potentially Inappropriate Medications Among Older Adults
Brief Title: An Intervention Study to Reduce the Use and Impact of Potentially Inappropriate Medications Among Older Adults
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study funding period reached conclusion. Sample size sufficient to complete the analysis on benzodiazepines.
Sponsor: Centre de Recherche de l'Institut Universitaire de Geriatrie de Montreal (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Cara Tannenbaum, Dr., Centre de Recherche de l'Institut Universitaire de Geriatrie de Montreal
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CIHR-2009MOP-201314-KTE
Record Dates: First submitted 2010-06-21; First posted 2010-06-22 (Estimated); Last update posted 2013-05-15 (Estimated); Status verified 2013-05

CONDITIONS: Polypharmacy; Incontinence; Insomnia; Anxiety
Keywords: Polypharmacy; Benzodiazepine use; Oxybutynin use; cognition disorders/drug therapy; incontinence
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Educational intervention (Experimental): Administration of an educational intervention to inform patients of the risks and safe alternatives to their current potentially inappropriate medication. The textual content of this knowledge transfer tool will be divided into three parts: a) presentation of the evidence-based risks associated with the targeted potentially inappropriate medication (e.g. benzodiazepines); b) presentation of evidence-based equally or more effective therapeutic substitutes for the medical condition (e.g. insomnia and anxiety); and c) presentation of evidence based tapering recommendations where applicable.
  Interventions: Behavioral: knowledge transfer tool
- Wait-list group (No Intervention)

INTERVENTIONS:
Behavioral: knowledge transfer tool — knowledge transfer tool for empowering patients to engage in collaborative discontinuation of potentially inappropriate medication with their pharmacist and/or physician
  Arms: Educational intervention

SUMMARY:
An educational intervention targeting community-dwelling older adults will lead to a reduction in potentially inappropriate prescriptions (e.g. benzodiazepines, oxybutynin).

Cessation of potentially inappropriate medications (e.g. benzodiazepines, oxybutynin)will lead to improved cognitive outcomes in older adults.

DETAILED DESCRIPTION:
This study tests the effectiveness of a knowledge transfer tool for empowering patients to engage in collaborative discontinuation of potentially inappropriate medication with their pharmacist and/or physician

ELIGIBILITY:
Inclusion Criteria:

* 65 year old human adults
* who fill a prescription for at least 5 medications
* community dwelling
* chronic use (3 months or longer) of at least one potentially inappropriate medication (e.g. benzodiazepine, oxybutynin)

Exclusion Criteria:

* patients with severe mental illness, dementia and epilepsy
* concomitant consumption of any other antipsychotic medication (including lithium, olanzapine, clozapine, quetiapine, risperidone, haloperidol etc.)
* concomitant consumption of any antiepileptic (including carbamazepine, valproate, gabapentin, lamotrigine, topiramate, oxcarbazepine etc.)
* concomitant consumption of a cholinesterase inhibitor or memantine

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 300 (Actual)
Dates: Start 2010-06; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Complete discontinuation of the targeted potentially inappropriate medication (e.g. benzodiazepines, oxybutynin) | 6 months post-intervention

SECONDARY OUTCOMES:
Cognitive function | 6-months post-intervention
  Montreal cognitive assessment instrument Rey's auditory verbal learning test (immediate memory, learning, and delayed recall)
Sleep efficiency | 6-months
  Sleep efficiency as documented with a sleep diary
incontinence-related self-efficacy | 6-months post-intervention
  incontinence-related self-efficacy as measured with the geriatric self-efficacy index
frequency of urinary incontinence episodes | 6-months post-intervention
  frequency of urinary incontinence as measured with a 72-hour bladder diary

CONTACTS AND LOCATIONS:
Overall Officials: Cara Tannenbaum, MD, Principal Investigator — Centre de recherche de l'Institut universitaire de gériatrie de Montréal
Locations (1):
- Le Groupe Jean Coutu Inc., Longueuil, Quebec, Canada

REFERENCES:
- [Derived] Martin P, Tannenbaum C. A realist evaluation of patients' decisions to deprescribe in the EMPOWER trial. BMJ Open. 2017 May 4;7(4):e015959. doi: 10.1136/bmjopen-2017-015959. PMID 28473524
- [Derived] Martin P, Tannenbaum C. Use of the EMPOWER brochure to deprescribe sedative-hypnotic drugs in older adults with mild cognitive impairment. BMC Geriatr. 2017 Jan 31;17(1):37. doi: 10.1186/s12877-017-0432-5. PMID 28143413
- [Derived] Tannenbaum C, Martin P, Tamblyn R, Benedetti A, Ahmed S. Reduction of inappropriate benzodiazepine prescriptions among older adults through direct patient education: the EMPOWER cluster randomized trial. JAMA Intern Med. 2014 Jun;174(6):890-8. doi: 10.1001/jamainternmed.2014.949. PMID 24733354
- [Derived] Martin P, Tamblyn R, Ahmed S, Tannenbaum C. An educational intervention to reduce the use of potentially inappropriate medications among older adults (EMPOWER study): protocol for a cluster randomized trial. Trials. 2013 Mar 20;14:80. doi: 10.1186/1745-6215-14-80. PMID 23514019